CLINICAL TRIAL: NCT01024140
Title: Open Trial of Escitalopram Treatment for Male Subjects With Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern California Institute of Research and Education (Other)
Responsible Party: Thomas C. Neylan, M.D., UCSF / VAMC / NCIRE
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEY-608
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Chronic Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Escitalopram; Efficacy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Escitalopram (Experimental): Flexible dose (5-20mg/day) of escitalopram monotherapy.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Subjects were started on 5mg escitalopram. Medication was increased as tolerated in weekly 2.5, 5 or 10 mg increments, until a maximally tolerated dosage or a clinical response was achieved. The final dosage ranged from 5 to 20 mg/day.
  Other Names: Lexapro

SUMMARY:
The primary aim of this pilot study is to test the efficacy of the selective serotonin re-uptake inhibitor, Escitalopram, in the treatment of posttraumatic stress disorder (PTSD) in an open clinical trial.

A secondary aim is to determine whether treatment with escitalopram increases plasma allopregnanolone levels in patients with PTSD and if increases in allopregnanolone levels are correlated with treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-IV TR PTSD and a score > 40 on the CAPS, as a result of a traumatic event that occurred at least 6 months prior to evaluation.

Exclusion Criteria:

* Lifetime history of bipolar or any psychiatric disorder with psychotic features.
* Prominent suicidal or homicidal ideation.
* History of alcohol abuse/dependence within the past 3 months.
* History of drug abuse/dependence within the past 6 months.
* Subjects who plan to start a new form of psychotherapy during the protocol.
* History of sleep apnea, neurological disorder and/or current systemic illness affecting central nervous system function.
* History of myocardial infarction in the past year.
* Subjects on antipsychotic medications, systemic steroid medication, antidepressants, mood stabilizers, antianxiety medication, or benzodiazepines within the past 2 weeks.
* Use of Citalopram or Escitalopram within the past 6 months.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2003-02; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The Clinician Administered PTSD Scale | Administered at baseline (prior to treatment) and week 12

SECONDARY OUTCOMES:
PTSD Checklist | Each Visit: Week 0, 2, 4, 6, 8, & 12
Beck Depression Inventory | Each Visit: Week 0, 2, 4, 6, 8, & 12
Profile of Mood State | Each Visit: Week 0, 2, 4, 6, 8, & 12
Social Adjustment Scale | Initial, Mid-Trial and Final Assessments
Quality of Life Inventory | Initial, Mid-Trial and Final Assessments

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Neylan, MD, Principal Investigator — UCSF / VAMC / NCIRE